CLINICAL TRIAL: NCT02514798
Title: Pilot Study of Physiological Effect of High-Flow Nasal Cannula on Respiratory Pattern and Work of Breathing in Severe COPD Patients
Brief Title: Pilot Study of Physiological Effect of High-Flow Nasal Cannula on Respiratory Pattern and Work of Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-11570
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: COPD
Keywords: COPD; HFNC; work of breathing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Gastric Balloon; Drug Delivery Systems; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-flow humidified nasal oxygen delivery system (Experimental): We will describe effects of varying settings of high-flow nasal oxygen (10-30-45-60 L/min) on respiratory rate, tidal volume, and diaphragmatic work of breathing in patients with severe COPD. We will also describe changes in gas exchange and effects on the subjects' comfort and dyspnea. This will be measured using, esophageal and gastric balloons, respiratory inductance plethysmography (RIP) system, and Sentec transcutaneous monitoring system.
  Interventions: Other: Esophageal and gastric balloons; Other: Respiratory Inductance Plethysmography (RIP) system; Other: Sentec transcutaneous monitoring system; Device: High-flow humidified nasal oxygen delivery system
- CPAP (Positive Control) (Active Comparator): We want to describe the breathing responses to varying setting of CPAP in the subject population. We plan to use the CPAP response as a "positive control", to determine if our population responds as described by CPAP studies in the literature. This will be measured using, esophageal and gastric balloons, respiratory inductance plethysmography (RIP) system, and Sentec transcutaneous monitoring system.
  Interventions: Other: Esophageal and gastric balloons; Other: Respiratory Inductance Plethysmography (RIP) system; Other: Sentec transcutaneous monitoring system; Device: CPAP (Positive Control)

INTERVENTIONS:
Other: Esophageal and gastric balloons — Esophageal and gastric pressures will be measured with an esophageal ballon positioned at the lower third of the esophagus, filled with 0.5 mL of air and a gastric balloon filled with 1 mL of air. The proper position of balloons will be verified using the occlusion test as previously described. Transdiaphragmatic pressure (Pdi) is calculated as the difference between gastric (Pga) and esophageal (Pes) pressure. The pressure time integrals of the diaphragm and the other inspiratory muscles are calculated per breath (PTPdi/b and PTPes/b, respectively) and per minute (PTPdi/min and PTPes/min). Measurements will be collected at baseline, at each randomized HFNC and CPAP settings during the last 4 minutes of each 10 minutes session.
Other: Respiratory Inductance Plethysmography (RIP) system — Inspiratory tidal volume (VTi), respiratory rate (RR), breath duration (Ttot), inspiratory time (Ti) and fractional inspiratory time (Ti/Ttot) will be determined using a Respiratory Inductive Plethysmography (RIP) system. This will measure the thoracic and abdominal excursion of the subjects via two inductive wires which are sewn into the elastic bands that encircle the thorax and abdomen. The acquired signals represent changes in cross-sectional area and, following calibration to determine the relative contribution of each signal, and volume calibration using spirometry, their weighted sum will reflect VTi. The RIP companion software will be used to derive RR, Ttot, Ti and Ti/Ttot on a breath by breath basis.
Other: Sentec transcutaneous monitoring system — The oxygenation, the level of carbon dioxide, and the heart rate will be recorded using the Sentec transcutaneous monitoring system: a probe will be placed at the earlobe or on the forehead, and it will measure in a noninvasive way these parameters.
Device: High-flow humidified nasal oxygen delivery system
  Arms: High-flow humidified nasal oxygen delivery system
Device: CPAP (Positive Control)
  Other Names: Continuous Positive Airway Pressure
  Arms: CPAP (Positive Control)

SUMMARY:
Patients affected with severe parenchymal pulmonary diseases, such as Chronic Obstructive Pulmonary Disease (COPD ), may experience dyspnea at rest due to increased work of breathing and reduced oxygenation. The delivery of high-flow humidified nasal oxygen (HFNC) has been shown to have a positive-end-expiratory pressure (PEEP) effect and is able to flush out CO2 from the upper airways, reducing dead space ventilation. Furthermore it has been proven to reduce the respiratory rate shortly after its initiation. These multiple actions offer the potential of changing the respiratory pattern and reducing work of breathing, improving the efficiency of breathing.

In this short-term, physiological, open, randomized, cross-over pilot study the investigator swill describe the effects of varying settings of high-flow nasal oxygen on respiratory rate, tidal volume, and diaphragmatic work of breathing in patients with severe COPD. The investigators will also describe changes in gas exchange and effects on the subjects' comfort and dyspnea and the breathing responses to varying setting of CPAP in the subject population.

DETAILED DESCRIPTION:
HFNC has been shown to have many advantages in the treatment of acutely hypoxemic patients, improving their clinical outcome. The exact mechanism underlying this beneficial effect is still not completely understood. Few studies have analyzed the effect of HFNC on ventilatory pattern and work of breathing. The majority of these studies have focused on the effects in healthy volunteers. Only one study from Braunlich et al. studied the effects of HFNC on COPD and interstitial lung disease (ILD) patients, showing that high-flow nasal oxygen reduces respiratory rate and increases the tidal volume in these patients.

In adults, a low flow range from 5 to 10 L/min is comparable to flow received by standard oxygen devices (nasal cannula or facial mask). Patients with underlying pulmonary diseases, as in our study population, have a higher inspiratory flow demands range (from 30 to 120 L/min during an acute respiratory failure episode) compared to healthy subjects.

We expect to observe physiological changes in our outcomes with the proposed Optiflow ™ settings of a minimal therapeutic flow of 30 L/min, intermediate of 45 L/min, and the maximal flow rate of 60 L/min. There is an extensive clinical experience using high flow rates in these ranges and they are generally very well tolerated. As mentioned above, HFNC generates a Positive End Expiratory Pressure (PEEP) comparable to CPAP range of 4 - 8 cmH2O (the minimal and the maximal PEEP generated by the HFNC).

Future studies, based on this pilot study, will differ from previous ones in the following ways:

1. We are testing a different technology. The Optiflow delivers substantially higher flow rates than in the previous Braunlich study13.That study used a single flow rate of 24 L/min whereas we are examining a range of flows that extend considerably higher (30 to 60L/min). We are interested in determining how the effects of higher flow rates compare to those in the range used in the Braunlich study, but we are not able to compare the devices directly because the latter device is not available in the US. It is important to understand whether there is any efficacy advantage to using the higher flow rates available with the Optiflow.
2. Future studies will aim to understand mechanisms of the effect of high flow nasal oxygen.

   1. Are the effects that we anticipate seeing related to changes in inspiratory muscle effort as determined by measurement of transdiaphragmatic pressure and calculation of the pressure time product of the diaphragm?
   2. Or does the flushing of dead space in the nasopharynx improve ventilatory efficiency so that gas exchange can remain stable or even improve (as determined by measurements of minute volume and transcutaneous PCO2 (PtcCO2)? This has implications for use of HFNC to treat patients with COPD exacerbations who are developing respiratory muscle fatigue.

1) Our focus will be on COPD patients for whom the use of HFNC has not been studied much to date. Most studies have focused on patients with hypoxemic respiratory failure. It is important to understand how HFNC affects breathing pattern and gas exchange in COPD patients because earlier reports suggest that excessive concentrations of oxygen administered to COPD patients retaining CO2 can actually worsen the CO2 retention by blunting respiratory drive. The reduction in respiratory rate and minute volume noted by Braunlich et al could represent a blunting effect of O2 on drive to breathe and could promote greater CO2 retention. By monitoring PCO2, something the Braunlich study didn't do, we can assess this possibility.

2) We wish to evaluate the effect of CPAP on the same breathing indices as with HFNC in our COPD patients. We plan to use the CPAP response as a "positive control", to determine if our population responds as described by CPAP studies in the literature. Prior studies have demonstrated that in patients with severe COPD, using CPAP in the range we are proposing, lowers the diaphragmatic work of breathing and we wish to determine if our population manifests a similar effect.

Thus future studies, based on the data obtained from this pilot study, will extend the Braunlich et al study by evaluating the effects of higher flow rates using a different technology available in the US, determining effects on inspiratory muscle effort, and monitoring gas exchange which is important from both mechanistic and safety perspectives. We hypothesize that the higher flow rates will have a greater blunting effect on breathing pattern than a low flow rate and that there will be an improvement in ventilator efficiency that will be associated with decreased breathing work of the diaphragm.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are 18 or more years of age
* Chronic respiratory failure, defined as indication for long-term oxygen therapy
* Underlying diagnosis of severe COPD (GOLD stage III or IV)

Exclusion Criteria:

* Recent (<1 month) exacerbation Acute exacerbation is defined as a sudden worsening of COPD symptoms (shortness of breath, quantity and color of phlegm) requiring a change in the baseline therapy.
* Respiratory rate at rest >28/min
* Subject requires > 6 L/min nasal O2 to maintain SpO2 >88% at rest
* Subject has severe dyspnea at rest
* Subject has swallowing disorder or chronic aspiration
* Prior esophageal surgery, known esophageal stricture or any other condition that would place the subject at risk during balloon placement
* Recent (< 1 month) abdominal and thoracic surgery
* Severe coagulopathy (defined as platelet count <5000/μL or international normalised ratio >4)
* Subject is too cognitively impaired to give subjective ratings for visual analogue scale.The PI and the Co-Investigators will assess the patient cognition using the Mini Mental State Examination (MMSE)
* Allergy or sensitivity to lidocaine
* Inability to obtain informed consent
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
respiratory rate | 90 minutes
  respiratory rate (RR) will be determined using a Respiratory Inductive Plethysmography (RIP) system. This will measure the thoracic and abdominal excursion of the subjects via two inductive wires which are sewn into the elastic bands that encircle the thorax and abdomen. The acquired signals represent changes in cross-sectional area and, following calibration to determine the relative contribution of each signal, and volume calibration using spirometry, their weighted sum will reflect VTi. The RIP companion software will be used to derive RR. It will be expressed as breaths per minute
tidal volume | 90 minutes
  Inspiratory tidal volume (VTi) will be determined using a Respiratory Inductive Plethysmography (RIP) system. This will measure the thoracic and abdominal excursion of the subjects via two inductive wires which are sewn into the elastic bands that encircle the thorax and abdomen. The acquired signals represent changes in cross-sectional area and, following calibration to determine the relative contribution of each signal, and volume calibration using spirometry, their weighted sum will reflect VTi (mL).
diaphragmatic work of breathing | 90 minutes
  Esophageal and gastric pressures will be measured with an esophageal ballon positioned at the lower third of the esophagus, filled with 0.5 mL of air and a gastric balloon filled with 1 mL of air. Transdiaphragmatic pressure (Pdi) is calculated as the difference between gastric (Pga) and esophageal (Pes) pressure. The pressure time integrals of the diaphragm and the other inspiratory muscles are calculated per breath (PTPdi/b and PTPes/b, respectively) and per minute (PTPdi/min and PTPes/min). Measurements will be collected at baseline, at each randomized HFNC and CPAP settings during the last 4 minutes of each 10 minutes session.

SECONDARY OUTCOMES:
changes in gas exchange | 90 minutes
  The oxygenation and the level of carbon dioxide will be recorded using the Sentec transcutaneous monitoring system: a probe will be placed at the earlobe or on the forehead, and it will measure in a noninvasive way these parameters.
effects on the subjects' comfort | 90 minutes
  Subject comfort during each setting will be evaluated using a Numeric rating scale (NRS). The subjects will be asked by the investigator to answer the following question: "How do you feel your comfort is at this moment?''. For each condition tested, the subject places a finger on the number that best represents their level of breathing comfort (from 0 to 10)
effects on the subjects' dyspnea | 90 minutes
  Subject breathing during each setting will be evaluated using a Numeric rating scale (NRS). The subjects will be asked by the investigator to answer the following question: "How do you feel your breathing is at this moment?''. For each condition tested, the subject places a finger on the number that best represents their level of breathing comfort (from 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hill, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dysart K, Miller TL, Wolfson MR, Shaffer TH. Research in high flow therapy: mechanisms of action. Respir Med. 2009 Oct;103(10):1400-5. doi: 10.1016/j.rmed.2009.04.007. Epub 2009 May 21. PMID 19467849
- [Background] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404
- [Background] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Background] El-Khatib MF. High-flow nasal cannula oxygen therapy during hypoxemic respiratory failure. Respir Care. 2012 Oct;57(10):1696-8. doi: 10.4187/respcare.02072. No abstract available. PMID 23013907
- [Background] Sztrymf B, Messika J, Bertrand F, Hurel D, Leon R, Dreyfuss D, Ricard JD. Beneficial effects of humidified high flow nasal oxygen in critical care patients: a prospective pilot study. Intensive Care Med. 2011 Nov;37(11):1780-6. doi: 10.1007/s00134-011-2354-6. Epub 2011 Sep 27. PMID 21946925
- [Background] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Background] Mundel T, Feng S, Tatkov S, Schneider H. Mechanisms of nasal high flow on ventilation during wakefulness and sleep. J Appl Physiol (1985). 2013 Apr;114(8):1058-65. doi: 10.1152/japplphysiol.01308.2012. Epub 2013 Feb 14. PMID 23412897
- [Background] Braunlich J, Beyer D, Mai D, Hammerschmidt S, Seyfarth HJ, Wirtz H. Effects of nasal high flow on ventilation in volunteers, COPD and idiopathic pulmonary fibrosis patients. Respiration. 2013;85(4):319-25. doi: 10.1159/000342027. Epub 2012 Nov 1. PMID 23128844
- [Background] Prinianakis G, Delmastro M, Carlucci A, Ceriana P, Nava S. Effect of varying the pressurisation rate during noninvasive pressure support ventilation. Eur Respir J. 2004 Feb;23(2):314-20. doi: 10.1183/09031936.03.00010203. PMID 14979510
- [Background] Vitacca M, Ambrosino N, Clini E, Porta R, Rampulla C, Lanini B, Nava S. Physiological response to pressure support ventilation delivered before and after extubation in patients not capable of totally spontaneous autonomous breathing. Am J Respir Crit Care Med. 2001 Aug 15;164(4):638-41. doi: 10.1164/ajrccm.164.4.2010046. PMID 11520729